CLINICAL TRIAL: NCT00647517
Title: Chung Shan Medical University Hospital, Taiwan
Brief Title: Tramadol/Acetaminophen(Ultracet) AS add-on Therapy in the Treatment of Patients With Ankylosing Spondylitis
Acronym: CS07102
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Cheng-Chung Wei, Chung Shan Medical University Hospital / Clinical trial center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: CSH-CMCTC-96-013
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2010-04-01 (Estimated); Status verified 2008-01

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Ultracet

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ultracet (Experimental)
  Interventions: Drug: Ultracet
- placebo (Placebo Comparator)
  Interventions: Drug: Ultracet

INTERVENTIONS:
Drug: Ultracet — For the treatment arm: Tramadol 37.5 mg/APAP 325 mg combination tablets (Ultracet®) one tablet twice a day plus aceclofenac tablet per oral 100 mg twice a day.
  For the control group: Placebo plus aceclofenac tablet per oral 100 mg twice a day.

SUMMARY:
Tramadol 37.5 mg/APAP 325 mg combination tablets (ULTRACET®) were effective and safe as addon therapy with COX-2 NSAID for treatment of osteoarthritis (5) and chronic low back pain (6).There is no clinical trial regarding tramadol usage in chronic inflammatory arthritis such as rheumatoid arthritis (RA) or ankylosing spondylitis. It would be important to do a pilot clinical trial on add-on effect of tramadol to NSAID in patients with AS or RA.

DETAILED DESCRIPTION:
Ankylosing spondylitis (AS) is a chronic inflammatory arthritis causing back pain, peripheral arthritis and enthesitis due to genetic background and autoimmunity. Patients with ankylosing spondylitis usually suffered from chronic pain over spine and peripheral joints since their second or third decades. It may also cause severe social and psychological burden to patients and their family.

Exercise and non-steroid anti-inflammatory drugs (NSAID) are the standard first-line treatments for AS（1）. Only 50% of patients with AS reach the ASAS response criteria（2） in clinical trials. Patients with severe disease activity should be put on disease-modifying anti-rheumatic drugs (DMARD), such as sulfasalazine（3） and anti-TNF biological agents. Add-on of acetaminophen and low dose anti-depressant （4）can slightly improve the response rate. However, there is no data if tramadol or ultracet can benefit AS.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of AS, as defined by Modified New York Criteria for Ankylosing Spondylitis
2. Active AS, defined by Bath ankylosing spondylitis disease activity index (BASDAI) >3 cm at screening visit.
3. Between 18 and 70 years of age.

Exclusion Criteria:

1. Change of dosage of disease modifying antirheumatic drugs (DMARDs) including glucocorticoid, hydroxychloroquine, sulphasalazine, and methotrexate within 4 weeks of baseline.
2. Change of dosage of biological agents within 4 weeks of baseline.
3. Abnormality in chemistry profiles: serum creatinine 3.0 mg/dl; alanine aminotransferase (ALT[SGPT]) 5 times the laboratory's upper limit of normal.
4. Pregnant or breast-feeding women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study is response defined by ASAS Response at 20% level at week 12. These criteria include measures of pain, function, inflammation, and patient global assessment of disease. | 1 year

SECONDARY OUTCOMES:
there is no secondary outcome. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: James WEI, MD, PhD., Principal Investigator — Department of rheumatology
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan